CLINICAL TRIAL: NCT03369470
Title: A New App Home Based Dexterity Training in Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: App Based Dexterity Training in Multiple Sclerosis
Acronym: AppDext
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Tim Vanbellingen, Head of department, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-00768
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Dexterity (Experimental)
  Interventions: Behavioral: App Dexterity
- Theraband (Active Comparator)
  Interventions: Behavioral: Theraband

INTERVENTIONS:
Behavioral: App Dexterity — App based dexterity training by means of Finger Zirkus (see for more details: www.fingers-in-motion.de)
  Arms: App Dexterity
Behavioral: Theraband — Active control being five traditional hand strengthening (Thera-band) exercises, which we published in our previous RCT, being feasible and effective in improving dexterity (for more details see for Kamm et al. 2015).
  Arms: Theraband

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system and the most common cause of non-traumatic disability in young adults (Kamm et al. 2014; Vanbellingen & Kamm, 2016). It is a heterogeneous disease, which is associated with long-term disability, leading to reduced quality of life (QoL). Disease-modifying pharmacological therapies (DMT) decrease activity and progression of the disease, and symptomatic pharmacological treatments reduce complaints to a certain extent, however MS patients often still suffer from various neurological deficits during the course of their disease (Kamm et al. 2014). Consequently, specific non-pharmacological therapies are needed in order to further reduce disability, eventually resulting in better QoL (Lamers et al. 2016; Vanbellingen & Kamm, 2016).

Impaired dexterity is a frequently observed impairment, affecting up to 76% of patients with MS (Johannson et al. 2007). The different neurological deficits caused by MS, such as ataxia, spasticity, sensory-motor deficits, and apraxia may be alone or in combination, impair manual dexterity (Kamm et al. 2012; Heldner, Vanbellingen et al. 2014). MS patients experience impairments in the performance of several activities of daily living (ADL), such as grooming, cooking, etc. Sometimes these problems are even associated with loss of work, and lack of social integration (Chruzander et al. 2013).

The effectiveness of the app based exercises still needs to be proven. With respect to dexterity, a first new app has been developed called "Finger Zirkus", by a team of experts including an occupational therapist, graphic designer, and IT expert. The app is already available to be downloaded from google play store or apple store (see for more details: www.fingers-in-motion.de).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for MS patients are as follows: males and females, age 18 to 75, diagnosis of MS (primary or secondary progressive, relapsing-remitting) following the McDonald criteria (Polman et al. 2011). In addition, patients must report difficulties in manual dexterity that impact ADL and/or have a pathological nine Hole Peg Test (9HPT) or Coin Rotation test (CRT) according to cut-off values (Mathiowetz et al. 1985; Heldner, Vanbellingen et al. 2014).

Exclusion Criteria:

* The exclusion criteria will be other conditions that may hand function or, impaired cognitive functioning (Mini Mental Status Examination score less than 24).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
AMSQ, Arm Function in Multiple Sclerosis Questionnaire (AMSQ) | 4 weeks
  AMSQ is a patient recorded outcome measurement for manual dexterity in MS patients (Mokkink et al. 2015).
  The "Arm Function in Multiple Sclerosis Questionnaire" (AMSQ) measures manual dexterity in patients with MS. It contains 31 questions on a unidimensional scale that are formulated as 'during the past two weeks, to what extent has MS limited your ability to ......?'. Response categories are from one to six ('not at all', 'a little', 'moderately', 'quite a lot', 'extremely', and 'no longer able to'). One final sum score is obtained with higher scores indicating more dexterous difficulties.The Dutch version showed good validity, test-retest reliability (ICC 0.90; SEM 5.6) and inter-observer reliability (ICC 0.95; SEM 7.2)

SECONDARY OUTCOMES:
Nine Hole Peg Test (9HPT) | 4 weeks
  9HPT is a reliable, valid and sensitive in detecting impaired dexterity in patients with MS (Lamers et al. 2014).
  The Nine Hole Peg Test (9HPT) is reliable (ICC values 0.80-0.99), valid and sensitive in detecting impaired dexterity in patients with MS. Patients were seated at a table with a shallow container holding nine pegs and a plastic block with nine empty holes. All pegs had to be put one at a time into the holes and then removed again one at a time into the shallow container. The time to complete the task was recorded twice on both hands and mean values were taken for each hand. If patients could not perform the CRT due to impaired manual dexterity, an arbitrarily chosen value of 300 seconds was chosen.
Multiple Sclerosis Impact Scale 29 (MSIS 29) | 4 weeks
  is a health-rated quality of life questionnaire (HRQoL) assessing the impact of MS on physical and psychological functions (Hobart et al. 2001).
  The Multiple Sclerosis Impact Scale (MSIS-29) is valid and reliable (ICC 0.80 - 0.87) in measuring the impact of MS on ADL.It contains 29 items comprising to a physical (MSIS-29 physical) and psychological impact scale (MSIS-29 psychological). All items are scored from 'not at all' to 'extremely' on a five-point Likert scale.
Coin Rotation Task (Kamm et al. 2012) | 4 weeks
  is a measure for dexterity. The Coin Rotation Task (CRT) has been validated in assessing manual dexterity in patients with MS. Patients had to rotate a 50 Swiss Rappen coin (corresponding to a dime or 2-cent Euro coin) as fast as possible between their thumb, index and middle finger. The time to perform 20 half turns was measured twice on both hands and mean values were taken for each hand. If patients could not perform the CRT due to impaired manual dexterity, an arbitrarily chosen value of 300 seconds was taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

REFERENCES:
- [Derived] van Beek JJW, Lehnick D, Pastore-Wapp M, Wapp S, Kamm CP, Nef T, Vanbellingen T. Tablet app-based dexterity training in multiple sclerosis (TAD-MS): a randomized controlled trial. Disabil Rehabil Assist Technol. 2024 Apr;19(3):889-899. doi: 10.1080/17483107.2022.2131915. Epub 2022 Oct 29. PMID 36308305